CLINICAL TRIAL: NCT03573024
Title: Safety and Efficacy of Venetoclax and Azacitidine for Newly Diagnosed Non-Elderly Adult Patients (Aged 18-59) With Acute Myeloid Leukemia
Brief Title: Venetoclax and Azacitidine for Non-Elderly Adult Patients With Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-0709.cc; NCI-2018-02119 (Other: CTRP)
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: Venetoclax; Azacitidine; Non-Elderly; Previously Untreated
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Azacitidine and Venetoclax (Experimental): Azacitidine will be given intravenously for 7 days. Venetoclax will be given orally. The patient will start out with 100mg and progress to 600mg. Once 600mg is reached, the patient will stay at this dose until the 28 day cycle is finished.
  Interventions: Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — On day 1 of cycle 1, azacitidine 75 mg/m2 SC or IV will be given, and will continue for 7 days.
Drug: Venetoclax — Starting on day 1 of cycle 1, venetoclax will be initiated. It will be dose escalated to a target dose of 600 mg in the following manner: 100 mg on day 1, 200 mg on day 2, 400 mg on day 3 and 600 mg on day 4. The patient then continues to take the 600mg dose for the remainder of the 28 day cycle. Each dose of venetoclax will be self-administered with approximately 240 mL of water within 30 minutes after the completion of a meal, preferably breakfast. The dose should be administered at the same time each day. On days the subject is given azacitidine, venetoclax must be given first.

SUMMARY:
This study aims to treat non-elderly adult patients, who were previously untreated for acute myeloid leukemia, using venetoclax and azacitidine.

DETAILED DESCRIPTION:
This is a phase II study that seeks to treat patients ages 18-59 who have acute myeloid leukemia but have never been treated before. It will use venetoclax and azacitidine, and patients can receive up to four cycles of this medication. Depending on the level of recovery, patients will either be forced to come off study or have the option to continue the medication, receive maintenance therapy, or pursue an allogeneic stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for study participation if he/she meets the following criteria within 28 days prior to the first day of therapy (bone marrow biopsy can be performed 28 days prior to the first day of therapy). Historical records are permitted per Investigator discretion.

1. Subject must have confirmation of non-APL and AML by WHO criteria45
2. Subject must have received no prior treatment for AML
3. Age ≥18 years, ≤59 years
4. Without clinical signs of active central nervous system disease
5. Subject must have an Eastern Cooperative Oncology Group (ECOG) Performance status of ≤2
6. Subject must have adequate renal function as demonstrated by a calculated creatinine clearance ≥ 30 mL/min; determined via urine collection for 24-hour creatinine clearance or by the Cockcroft Gault formula
7. Subject must have adequate liver function as demonstrated by:

   * aspartate aminotransferase (AST) ≤ 3.0 × ULN*
   * alanine aminotransferase (ALT) ≤ 3.0 × ULN*
   * bilirubin ≤ 3.0 × ULN, unless due to Gilbert's syndrome* * Unless considered due to leukemic organ involvement
8. Non-sterile male subjects must use contraceptive methods with partner(s) prior to beginning study drug administration and continuing up to 90 days after the last dose of study drug. Male subjects must agree to refrain from sperm donation from initial study drug administration until 90 days after the last dose of study drug.
9. Female subjects who are pre-menopausal and have not had a hysterectomy or oophorectomy must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting therapy; 2) throughout the entire duration of treatment; 3) during dose interruptions; and 4) for at least 90 days after discontinuation of therapy (last dose of study drug).
10. Subject must voluntarily sign and date an informed consent, approved by an Institutional Review Board (IRB), prior to the initiation of any research directed screening procedures.
11. Subject must have adverse risk disease as defined by the European LeukemiaNet46 (Appendix B) 5.3.2 Exclusion Criteria

A subject will not be eligible for study participation if he/she meets any of the following criteria:

1. Subject has received disease modifying treatment for myelodysplastic syndrome (MDS) or AML. ATRA given for clinical suspicion of APL will not be exclusionary and no washout will be required in this scenario.
2. Subject is known to be positive for HIV. HIV testing is not required.
3. Subject is known to be positive for hepatitis B or C infection with the exception of those with an undetectable viral load. Hepatitis B or C testing is not required and subjects with serologic evidence of prior vaccination to HBV (i.e., HBs Ag-, anti-HBs+ and anti-HBc-) may participate
4. Subject has received within 7 days prior to the first dose of study drug:steroid therapy for anti-neoplastic intent; strong and moderate CYP3A inhibitors; strong and moderate CYP3A inducers.
5. Subject is informed that consumption of the following fruits is prohibited 3 days prior to the initiation of study treatment and throughout participation: grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Star fruit.
6. Subject has any history of clinically significant condition(s) that in the opinion of the investigator would adversely affect his/her participating in this study including, but not limited to:

   * New York Heart Association heart failure > class 2
   * Renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, or bleeding disorder independent of leukemia
7. Subject has a malabsorption syndrome or other condition that precludes enteral route of administration
8. Subject exhibits evidence of uncontrolled systemic infection requiring therapy (viral, bacterial or fungal)
9. Subject has a history of other malignancies prior to study entry, with the exception of:

   * Adequately treated in situ carcinoma of the breast or cervix uteri
   * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin
   * Prostate cancer with no plans for therapy of any kind
   * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
10. Subject has a white blood cell count >25 × 10^9/L or absolute blast count of >50 10^9/L. Hydroxyurea and leukapheresis are permitted, if clinically indicated.
11. Patients willing to receive intensive induction chemotherapy
12. Pregnant and breastfeeding females.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Response Rate, measured by the European Leukemia Net definition: (CRMRD-+CR+CRi+MLFS) | Study start date to study end date, or death, whichever comes first, up to 4 years
  The (CRMRD-+CR+CRi+MLFS) shows non-inferiority of venetoclax with azacitidine when compared with historical controls who received induction chemotherapy.

SECONDARY OUTCOMES:
Incidence of Minimal Residual Disease (MRD) Negative Responses | Study start date to study end date, or death, whichever comes first, up to 4 years
  Number of new cases of Complete Remission, Complete Remission with Incomplete Blood Count Recovery, or Morphologic Leukemia Free State. This will be measure by multi-dimensional flow cytometry with a sensitivity to 0.1%.
Remission Duration | Study start date to study end date, or death, whichever comes first, up to 4 years
  Remission Duration will be defined as the length of time a patient does not display leukemic blasts or extramedullary disease
One Year Event Free Survival | Study start date to study end date, or death, whichever comes first, up to 4 years
  Determined using Kaplan Meier survival analysis methods with 95% confidence intervals.
Overall Survival | Study start date to study end date, or death, whichever comes first, up to 4 years
  Overall Survival will be defined as the time from administration of the initial doses until death from any cause. Determined using Kaplan Meier survival analysis methods with 95% confidence intervals.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Study start date to study end date, or death, whichever comes first, up to 4 years
  Safety and tolerability analysis of azacitidine and venetoclax will be summarized by dose and severity as assessed by the Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0 and relationship to study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pollyea, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Universtiy of Colorado Hospital, Aurora, Colorado, United States